CLINICAL TRIAL: NCT00910221
Title: A Phase II Randomised, Double-blind, Placebo-controlled Study of the Effect of Atorvastatin on Postoperative Renal Function in Patients Undergoing Elective Cardiopulmonary Bypass.
Brief Title: Cardiopulmonary-bypass and Reno-protective Effect of Atorvastatin Trial
Acronym: CREAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Director of ICU research, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H2007/02810
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2009-08

CONDITIONS: Acute Kidney Dysfunction
Keywords: Cardiac surgery; Cardiopulmonary bypass; Oxidative stress; Acute renal dysfunction; Atorvastatin
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin tablet
  Arms: 1
Drug: Placebo — Placebo tablet
  Arms: 2

SUMMARY:
Acute kidney dysfunction is common after cardiac surgery. While many patients suffer no long-term ill effects from post-operative kidney dysfunction, some require initiation of dialysis therapy that can contribute to long-term morbidity. Further, there is evidence to suggest that those patients requiring dialysis after cardiac surgery have a higher risk of death in hospital.

The exact reasons why some patients develop acute kidney dysfunction after cardiac surgery is not well understood. However, research evidence to date has suggested that the presence of co-morbid illnesses (i.e., diabetes mellitus) and exposure to cardiopulmonary bypass (heart-lung machine used during operation when heart is stopped). Cardiopulmonary bypass, in particular, has been shown to over-activate several aspect of the body's immune system. Such over-activity can induce oxidative stress and contribute to acute kidney dysfunction.

The investigators believe that the statin drug, atorvastatin, might reduce the oxidative stress that occurs during cardiopulmonary bypass, and thus, prevent or reduce the magnitude of acute kidney dysfunction in those patients at highest risk. The investigators hope to give atorvastatin (40 mg orally) to patients immediately prior to and for 3 days after cardiac surgery, and to compare the effects on kidney function with patients who have not had atorvastatin.

Atorvastatin is the most commonly prescribed medication in Australia and is used to reduce blood cholesterol levels and decrease the risk of heart attacks and stroke. Recently, however, it has been discovered that atorvastatin may be useful for prevention of inflammation and oxidative stress in other conditions, such as following cardiac surgery with cardiopulmonary bypass.

Thus, the investigators plan to examine whether atorvastatin can prevent acute kidney dysfunction. This trial as planned is a pilot study. If atorvastatin shows promising evidence of reduction in acute kidney dysfunction, further studies on a larger scale would be required to justify its general use.

The investigators plan to determine whether atorvastatin, a statin drug, possesses kidney protective effects in patients at risk for perioperative acute kidney dysfunction after cardiac surgery and exposure to cardiopulmonary bypass.

This is a pilot, randomized, blinded, placebo-controlled trial.

The investigators plan to administer atorvastatin (40 mg orally) or placebo to patients immediately prior to and for 3 days after cardiac surgery. The atorvastatin/placebo will be given orally either by orogastric tube after induction of anaesthesia or swallowed by the patients.

Whether a particular patient receives the atorvastatin or placebo will be decided at random, and neither the patient nor the investigators will be aware of the allocated treatment.

The investigators plan to measure kidney function before and after cardiac surgery using the standard blood tests. The investigators also plan to measure markers of inflammation and oxidative stress in the blood. This may give insight into the mechanisms whereby atorvastatin exerts its effects. The investigators will also take four 20 ml samples of blood, spaced before, and after the operation, from the arterial catheter routinely inserted in every patient undergoing cardiac surgery.

The investigators believe that there will be no significant additional risk to a patient who participates in the study, and no discomfort other than that normally associated with cardiac surgery. Informed consent will be obtained from the patient prior to the operation by one of the investigators or the ICU research nurse. The clinical care of a patient who does not consent for any reason will not be affected.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical patients in whom the use of cardiopulmonary bypass was planned
* Written informed consent of patient
* Age > 18 years
* And having at least one ore more of the following risk factors for postoperative AKI:

  * Age =/> 70 years
  * Preoperative plasma creatinine >120 µmol/L, New York Heart Association class III/IV or LVEF <35%
  * Insulin dependent diabetes mellitus
  * Valve surgery (with or without coronary artery bypass graft)
  * Redo cardiac surgery

Exclusion Criteria:

* An emergency operation is indicated (within 24 hours after hospital admission or on intra-aortic balloon pump)
* Pregnancy is confirmed or breastfeeding is present
* A renal allograft is present
* Preoperative acute renal failure within 6 weeks (acute rise in serum creatinine > 50% from baseline) is present
* Pre-operative end stage renal disease (serum creatinine > 300 µmol/L) is present
* Chronic moderate to high dose corticosteroid therapy (>10 mg/d prednisone or equivalent) is present
* Known Allergy to Atorvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2010-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in serum creatinine from baseline to peak level | within first two-seven postoperative days

SECONDARY OUTCOMES:
Proportion of patients developing an increase in serum creatinine > 25% or >44µmicromol/L from baseline to peak level | within first two-seven postoperative days
Proportion of patients developing any of the RIFLE criteria: R, I or F | within first seven postoperative days
Proportion of patients developing any of the AKI stages: 1, 2 or 3 (using network definition) | within first seven postoperative days
Change in NGAL from baseline to peak | within first 24 postoperatively
Requirement of renal replacement therapy | within hospital stay
Length of stay in Intensive care | from admission to discharge from Intensive care
Length of stay in Hospital | from admission to discharge from hospital
Hospital-Mortality | during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Prowle JR, Calzavacca P, Licari E, Ligabo EV, Echeverri JE, Haase M, Haase-Fielitz A, Bagshaw SM, Devarajan P, Bellomo R. Pilot double-blind, randomized controlled trial of short-term atorvastatin for prevention of acute kidney injury after cardiac surgery. Nephrology (Carlton). 2012 Mar;17(3):215-24. doi: 10.1111/j.1440-1797.2011.01546.x. PMID 22117606